CLINICAL TRIAL: NCT02088515
Title: Nedaplatin (Jiebaishu®) and Docetaxel in Comparison With Cisplatin and Docetaxel Regimen for the First Line Treatment of Advanced Squamous Cell Carcinoma of Lung(IIIB/IV): Randomized, Controlled, Multicentre Study
Brief Title: Nedaplatin (Jiebaishu®) Combined With Docetaxel for Advanced Lung Squamous Cell Carcinoma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jiangsu Simcere Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5501068
Record Dates: First submitted 2014-03-06; First posted 2014-03-17 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2016-04

CONDITIONS: Squamous Cell Carcinoma
Keywords: Nedaplatin; lung squamous cell carcinoma
MeSH Terms: conditions — Carcinoma, Squamous Cell | interventions — nedaplatin; Cisplatin; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- experimental group (Experimental): experimental group: Nedaplatin(（80 mg/m2, i.v Day1）in combination with Docetaxel（75 mg/m2, i.v Day1）for each cycle, 4 cycles in total.
  Interventions: Drug: Nedaplatin; Drug: Docetaxel
- comparative group (Active Comparator): comparative group:Cisplatin (（75 mg/m2, i.v Day1 or 25 mg/m2 Day1-3）in combination with Docetaxel（75 mg/m2, i.v Day1）for each cycle, 4 cycles in total
  Interventions: Drug: Cisplatin; Drug: Docetaxel

INTERVENTIONS:
Drug: Nedaplatin
  Arms: experimental group
Drug: Cisplatin
  Arms: comparative group
Drug: Docetaxel

SUMMARY:
The treatment of squamous cell carcinoma of lung has not improved suffuciently. Nedaplatin is a second-generation platinum compound that is more active against squamous cell carcinoma of the lung with a response rate of 60%, issued by the finished Phase II trial in Japan.

ELIGIBILITY:
Inclusion Criteria:

1. primary lung squamous carcinoma confirmed by cytology and histology, excluding sputum examination.
2. IIIB-no radiotherapy indication /IV phased by ASLC 2009 TNM criteria.
3. at least one measurable tumor based on RECIST ( longest diameter: ≥20 mm by CT scan or 10 mm by spiral CT )
4. male or female, age≥18 or ≤75 years old
5. ECOG PS: 0 or 1
6. estimated time of survival: ≥12 weeks
7. suitable hematologic function: ANC≥2×109/L, PLC≥100×109/L and Hb≥9 g/dL
8. suitable liver function: Total bilirubin≤normal ULN, AST and ALT≤2.5×normal ULN, ALP≤5×normal ULN.
9. suitable renal function: Cr≤normal ULN,or Ccr≥60 ml/min
10. no history of chemotherapy
11. at the enrollment, the past operation has been over 4 weeks and the subject recovered.
12. for the female subject with the intact uterus, if amenorrhea is less than 24 months, pregnancy test must be negative within 28 days of enrollment. If pregnancy test has been past 7 days at the time of initial chemotherapy, urine pregnancy test must be done.
13. the authorized ICF must be signed

Exclusion Criteria:

1. having the other cancer in the recent five years, cured skin basal cell carcinoma and cervical carcinoma excluded.
2. having the evidence of CNS metastasis, no matter if treated; if being suspicious of CNS metastasis, CNS MRI or enhanced CT scan must be done within 28 days of enrollment.
3. AST and /or ALT>2.5×normal ULN, and ALP>5×normal ULN.
4. radiotherapy in the past (excluding palliative radiotherapy for pain relief and the measurable tumor outside the radio field)
5. chemotherapy in the past (excluding bisphosphonates )
6. having the other uncontrolled diseases.
7. the female in pregnancy or feeding.
8. the subjects with the productivity capacity, but refusal to use the effective contraception measure.
9. participating in other clinical trial and at the time of treatment period.
10. allergy to the tested drugs
11. having the other uncontrolled diseases
12. BMT had been done.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 290 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
progress free survival | 9 months
  after being enrolled, the subjects will be subject to 4 cycles chemotherapy (each cycle: 21 days). if complete response/partial response/stable desease is confirmed, the subjects will be followed up till to the sixth months.

SECONDARY OUTCOMES:
Objective Response Rate | 3 months
  the effectiveness will be evaluated after 2 cycles of chemotherapy is finished. 4 cycles of chemotherapy is needed for each subject.

OTHER OUTCOMES:
Adverse Events | 10 months
  Adverse Events will be recorded and monitored till to normal or basal level achieved.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hunan Xiangya Hospital, Changsha, Hunan
  - Nanjing Military General Hospital, Nanjing, Jiangsu
  - Shanghai Chest hospital, Shanghai, Shanghai Municipality
  - Xijing Hospital, Xian, Shanxi

REFERENCES:
- [Derived] Lu S, Chen Z, Hu C, Zhang J, Chen Y, Song Y, Zhao Q, Fan Y, Wu G, Ma Z, Fang J, Yu Q, Liu Z. Nedaplatin Plus Docetaxel Versus Cisplatin Plus Docetaxel as First-Line Chemotherapy for Advanced Squamous Cell Carcinoma of the Lung - A Multicenter, Open-label, Randomized, Phase III Trial. J Thorac Oncol. 2018 Nov;13(11):1743-1749. doi: 10.1016/j.jtho.2018.07.006. Epub 2018 Jul 11. PMID 30017831